CLINICAL TRIAL: NCT04019457
Title: Cereals and Intestinal Function: Investigations in Healthy Participants
Brief Title: Cereals and Intestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna19
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Endotoxemia; Diet, Healthy
MeSH Terms: conditions — Endotoxemia | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary fiber 1 (Experimental): Participants receive cereal flakes 1 to include it in their normal diet.
  Interventions: Other: Dietary intervention
- Dietary fiber 2 (Experimental): Participants receive cereal flakes 2 to include it in their normal diet.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Dietary intervention: Participants receive dietary fibers for a defined number of days.

SUMMARY:
The aim of the present study is to determine the effect of dietary fiber on intestinal function in healthy subjects.

DETAILED DESCRIPTION:
In the intervention study normal weight participants will receive defined amounts of different cereal flakes for several days. Before and after intervention parameters of intestinal function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI <25 kg/m2
* daily alcohol consumption <20g (men) or <10g (women)

Exclusion Criteria:

* food allergies or intolerances
* instable body weight
* BMI <18,5 kg/m2 or >25 kg/m2
* bariatric surgery within the last 5 years
* intake of antibiotics within the last month or during the study
* daily alcohol consumption >20g (men) or >10g (women)
* pregnancy and/or lactation period
* viral or bacterial infection during the last three weeks
* increased inflammatory markers of unknown reason
* chronic or acute disease of gastrointestinal tract

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in parameters of intestinal barrier function | 1 week
  Changes in endotoxin plasma levels

SECONDARY OUTCOMES:
Changes in blood lipid levels | 1 week
  Changes in triglyceride levels (mg/dl), changes in cholesterol levels (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No